CLINICAL TRIAL: NCT03834285
Title: EASL: European Registry of Liver Disease in Pregnancy
Brief Title: Liver Disease in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: European Association for the Study of the Liver (Unknown)
Responsible Party: Sponsor
Other Study IDs: 238575
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Pregnancy Disease; Cirrhosis, Liver; HELLP Syndrome; AFLP - Acute Fatty Liver of Pregnancy; Intrahepatic Cholestasis of Pregnancy
MeSH Terms: conditions — Liver Cirrhosis; HELLP Syndrome; Acute fatty liver of pregnancy; Intrahepatic Cholestasis of Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cirrhosis in pregnancy: Cirrhotic patients with a confirmed pregnancy will be placed into Cohort 1.
- Pregnancy-associated liver diseases: Patients who develop Acute Fatty Liver of Pregnancy, HELLP Syndrome / Intrahepatic Cholestasis of pregnancy will be placed into Cohort 2.

SUMMARY:
Liver Diseases in pregnancy represents rare disorders and current data is derived primarily from single centres and retrospective cohorts. Moreover, the population prevalence of these diseases is low and to-date, it has proven difficult to generate reliable data at a patient level.

This is a multi-center, prospective cohort study that will open at 3 centers within the UK; and 4 centers in the European Union. The investigators will aim to collect data and blood samples at various time points, for patients presenting with liver disease during pregnancy. The main rationale behind this study is to establish a platform that enables detailed review of the outcomes of these rare diseases; to help classify and stratify patients according to risk and develop interventional studies and care pathways to improve overall outcome.

DETAILED DESCRIPTION:
The objectives of the study are as follows:

Primary Objective:

To determine the characteristic physiological and biological changes exhibited by females who develop the following liver diseases during pregnancy.

* Acute fatty liver of pregnancy
* Severe cholestasis of pregnancy
* Severe HELLP syndrome/hypertensive disease
* Pre-existing cirrhosis and pregnancy This will be determined through analysis of the standard of care imaging (Liver Ultrasound and Transient Elastography) and blood results (liver function tests, white blood cells, platelets and scoring systems for assessing the severity of liver disease (ALBI, APRI, FIB4 and ELF scores). These results will be analysed over the course of the participant's pregnancy and again at delivery, to explore any particularly distinguishing parameter changes for each disease group.

Secondary Objectives

1. To determine the change in the reported quality of life of these participants either from diagnosis of pregnancy-associated liver disease or confirmation of pregnancy for pre-existing cirrhotic patients - up to 3 months' post-delivery.
2. To determine the mitochondrial DNA content of blood from patients with Acute Fatty Liver of Pregnancy.
3. Create an associated pan-European bio-resource (whole blood and serum) collection, which will offer an opportunity for ongoing collaborative translational research. Each participant will be given the option of donating additional research samples (15ml) of blood at each visit under the study for the bio-resource.

Data from cirrhotic patients will be collected from pre-pregnancy and during the first, second and third trimesters as well as at delivery and post-partum. Data from patients with AFLP/HELLP/ICP will be collected from pre-diagnosis, at first presentation of liver disease, at peak of liver disease, during the recovery period from peak liver disease as well as at delivery and post-partum.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients older than 18 years of age, willing and able to sign written informed consent.
2. Pregnant and presenting with any one of the following conditions (confirmed by local diagnosis):

   * Acute fatty liver of pregnancy
   * Severe cholestasis of pregnancy
   * Severe HELLP syndrome /hypertensive disease
   * Pre-existing cirrhosis and pregnancy
3. Able to provide written informed consent
4. Willing to provide access to records to necessary data can be collected.
5. Willing to complete additional quality of life questionnaires as per protocol.
6. Willing to consider donation of optional blood samples as per protocol.

Exclusion Criteria:

1. Unable to provide written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy study, so all participants must be female.
Study Population: Liver Diseases in pregnancy represent rare disorders and the numbers of patients affected in the overall population is low and therefore, it has proven difficult to generate reliable data. For example, the numbers of patients affected with these conditions in Europe are as follows:
  * Acute Fatty Liver affects 1:20,000 pregnant women
  * Severe Cholestasis - 1:3,000 pregnant women
  * Severe haemolysis, elevated liver enzymes and low platelets (HELLP syndrome) requiring transfer to a liver transplant centre or specialised hepatopancreatobiliary(HPB) centre at best estimate represents less than 0.01% of pregnancies.
  Patients with pre-existing cirrhosis and pregnancy represent approximately 0.003% of pregnancies, yet, to-date, less than 5 reliable publications exist in the literature to inform patient management.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2024-04-08 (Estimated); Study Completion 2025-04-08 (Estimated)

PRIMARY OUTCOMES:
Overall maternal and fetal health during pregnancy and post-delivery in females with liver disease | Data to be collected from pre-pregnancy to 3 months post-delivery
  Data from 100 patients will be collected across the EU who have either pre-exisiting cirrhosis or one of the three pregnancy-associated liver diseases that are to be studied in this protocol (AFLP, HELLP, ICP)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Heneghan, Study Chair — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No